CLINICAL TRIAL: NCT00738504
Title: INTENSIVE INSULIN THERAPY REALLY REDUCES THE INCIDENCE OF ACUTE KIDNEY INJURY IN CRITICALLY ILL PATIENTS? An Analysis Using the RIFLE Criteria for Definition of Acute Kidney Injury.
Brief Title: Intensive Insulin Therapy and Acute Kidney Injury. Analysis Using RIFLE Criteria.
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: JOSÉ RAIMUNDO ARAUJO DE AZEVEDO, HOSPITAL SAO DOMINGOS
Other Study IDs: HSaoDomingos N 051/2008
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Kidney; Injury
Keywords: Intensive insulin therapy; Carbohydrate restrictive strategy; RIFLE Criteria; Acute Kidney Injury; Critically ill patients; Acute
MeSH Terms: conditions — Wounds and Injuries; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1
- 2
- Group 1: Group 1 (Carbohydrate Restrictive Strategy). Patients received intravenous hydration with a glucose free solution (Ringer III) and enteral nutritional formula containing 33.3% carbohydrates, 16,7% proteins and 50% lipids (Glucerna, Abbott Laboratories). These patients received regular insulin subcutaneously four times daily, aiming to maintain blood glucose levels at least below 180 mg/dl, and, in stable patients, ideally below 150 mg/dl.
- Group 2: Group 2 (Intensive Insulin Therapy). Continuous intravenous insulin infusion was adjusted to maintain glycemic levels at least below 150 mg/dl, and, in stable patients and ideally, between 80 to 120 mg/dl. Patients were submitted to capillary glycemic measurements every 2 hours. The insulin dose was adjusted according to an algorithm run by nurses and overseen by physicians. These patients received glucosaline (5% glucose + 0.9 NaCl) hydration and enteral nutrition with a formula containing 45% carbohydrates, 17% proteins and 38% lipids (Diason, Nutricia Clinical Care Ltd).

SUMMARY:
The purpose of this study is to determine if intensive insulin therapy really reduces the incidence of acute kidney injury in critically ill patients, using for analysis the RIFLE criteria for definition of AKI.

ELIGIBILITY:
Inclusion Criteria:

* We included 337 adult patients, non pregnant, admitted from July 1, 2004 to December 31, 2006, to a 20-bed multidisciplinary ICU of a general hospital and to an 11-bed trauma center ICU that had at least two blood glucose levels above 150 mg/dl from three measurements obtained in the first 12 hours after admission.

Exclusion Criteria:

* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are going to evaluate retrospectively the occurrence of acute kidney injury defined by the RIFLE criteria in a population of patients submitted to two different strategies for glycemic control: a carbohydrate restrictive strategy or intensive insulin therapy. The protocol of the original trial that we are going to summarize below, was approved by the Research Ethical Committee of the Federal University of Maranhão. We included 337 adult patients, non pregnant, admitted from July 1, 2004 to December 31, 2006, to a 20-bed multidisciplinary ICU of a general hospital and to an 11-bed trauma center ICU that had at least two blood glucose levels above 150 mg/dl from three measurements obtained in the first 12 hours after admission.
Sampling Method: Probability Sample
Enrollment: 337
Dates: Start 2008-06

PRIMARY OUTCOMES:
To compare the renal function outcome, defined by the RIFLE criteria in patients submitted to two different regimens of glycemic control: a carbohydrate restrictive strategy and intensive insulin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, MD, Principal Investigator — Director. BRAZILIAN ASSOCIATION OF INTENSIVE CARE MEDICINE
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil